CLINICAL TRIAL: NCT02654132
Title: An Open Label, Randomized Phase 2 Trial of Pomalidomide/Dexamethasone With or Without Elotuzumab in Relapsed and Refractory Multiple Myeloma (ELOQUENT-3)
Brief Title: An Investigational Immuno-therapy Trial of Pomalidomide and Low-dose Dexamethasone With or Without Elotuzumab to Treat Refractory and Relapsed and Refractory Multiple Myeloma (ELOQUENT-3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Celgene (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-125; 2014-003282-19 (EudraCT Number)
Record Dates: First submitted 2015-12-31; First posted 2016-01-13 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elotuzumab Arm (Experimental): Biological:Elotuzumab (BMS-901608; HuLuc63)
  * Solution, Intravenous(IV),10 mg/kg(Cycles 1 and 2 weekly, on Days 1,8,15,22)
  * Solution, Intravenous(IV),20 mg/kg(Cycle 3 and Beyond: Day 1)
  Drug: Pomalidomide
  •Capsules,Oral,4 mg,once daily, on Days 1-21
  Other Name: Pomalyst
  Drug: Dexamethasone
  * Subjects ≤ 75 years old:
    •Tablets, Oral,28 mg, once daily on: Days 1,8,15,22(Cycles 1&2) Day 1(Cycle 3 and Beyond)
    •Solution, Intravenous(IV), 8 mg, once daily on: Days 1,8,15,22(Cycles 1&2) Day 1(Cycle 3 and Beyond)
    •Tablets, Oral,40 mg, once daily on: Days 8,15,22(Cycle 3 and Beyond)
  * Subjects > 75 years old:
    •Tablets, Oral,8 mg, once daily on: Days 1,8,15,22(Cycles 1&2) Day 1(Cycle 3 and Beyond)
    •Solution, Intravenous(IV), 8 mg, once daily on: Days 1,8,15,22(Cycles 1&2) Day 1(Cycle 3 and Beyond)
    •Tablets, Oral, 20 mg, once daily on: Days 8,15,22(Cycle 3 and Beyond)
  Other Names:
  Decadron,Dexamethasone ,Intensol,Dexpak,Taperpak
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone
- Control Arm (Active Comparator): Drug: Pomalidomide
  • Capsules, Oral, 4 mg, once daily, on Days 1-21 Other Name: Pomalyst
  Drug: Dexamethasone
  Subjects ≤ 75 years old:
  • Tablets, Oral, 40 mg, weekly on Days 1, 8, 15 and 22
  Subjects > 75 years old:
  • Tablets, Oral, 20 mg, weekly on Days 1, 8, 15 and 22,
  Other Names:
  * Decadron
  * Dexamethasone Intensol
  * Dexpak
  * Taperpak
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab
  Arms: Elotuzumab Arm
Drug: Pomalidomide
  Other Names: Pomalyst
Drug: Dexamethasone
  Other Names: Decadron, Dexamethasone, Intensol, Dexpak, Taperpak

SUMMARY:
The purpose of this study is to determine if adding Elotuzumab to Pomalidomide and low-dose dexamethasone is a more effective treatment of relapsed and refractory multiple myeloma compared to pomalidomide and low-dose dexamethasone by itself.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* ≥ 2 prior lines of therapy which must have included at least 2 consecutive cycles of lenalidomide and a proteosome inhibitor alone or in combination
* Documented refractory or relapsed and refractory multiple myeloma
* Refractory to proteosome inhibitor and lenalidomide, and to last treatment
* Relapsed and refractory patients must have achieved at least a partial response to previous treatment with proteosome inhibitor or lenalidomide, or both, but progressed within 6 months, and were refractory to their last treatment
* Measurable disease at screening
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Active plasma cell leukemia
* Prior treatment with pomalidomide
* Unable to tolerate thromboembolic prophylaxis while on the study
* Prior autologous stem cell transplant within 12 weeks
* Known Human Immunodeficiency Virus (HIV) infection or active hepatitis A, B, or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (55):
- United States (12):
  - Winship Cancer Institute, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - Beth Israel Comprehensive Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Rochester General Hospital, Rochester, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Va Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - St Francis Hospital, Greenville, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Northern Utah Associates, Ogden, Utah
  - University Of Washington, Seattle, Washington
- Local Institution, South Brisbane, Queensland, Australia
- Canada (3):
  - Local Institution, London, Ontario
  - CISSS de l'Outaouais, Gatineau, Quebec
  - Local Institution - 0048, Montreal, Quebec
- France (5):
  - Local Institution - 0022, Nantes
  - Local Institution - 0021, Paris
  - Local Institution - 0020, Pessac
  - Local Institution - 0019, Poitiers
  - Local Institution, Saint-Pierre
- Germany (7):
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - St. Barbara-Klinik, Hamm
  - Local Institution - 0041, Heidelberg
  - Local Institution - 0056, Kiel
  - Klinikum Der Johannes Gutenberg Universitaet Mainz, Mainz
  - Universitaetsklinikum Tuebingen, Tübingen
- Greece (2):
  - Laiko University Hospital, Athens
  - Alexandra General Hospital Of Athens, Athens
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Di Ancona, Ancona
  - A. O. U. Di Bologna, Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Local Institution, Roma
  - Universita' La Sapienza, Roma
  - Azienda Ospedaliera Citta' Della Salute E Della Scienza Di Torino, Torino
- Japan (8):
  - Local Institution - 0030, Nagoya, Aichi-ken
  - Local Institution - 0069, Morioka, Iwate
  - Local Institution - 0031, Kyoto, Kyoto
  - Local Institution - 0029, Niigata, Niigata
  - Local Institution - 0027, Shibuya-ku, Tokyo
  - Local Institution - 0028, Tachikawa-shi, Tokyo
  - Local Institution - 0067, Kasama-shi
  - Local Institution - 0032, Okayama
- Netherlands (4):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Maastrict
  - Local Institution, Utrecht
- Poland (3):
  - Oddzial Kliniczny Hematologii i Profilaktyki Chorob Nowotworowych, Chorzów
  - Local Institution, Lublin
  - Oddzial Hematologii i Transplantacji Szpiku, Poznan
- Spain (4):
  - Local Institution, Pamplona, Navarre
  - Local Institution, Barcelona
  - Local Institution - 0024, Madrid
  - Local Institution, Valencia

REFERENCES:
- [Derived] Dimopoulos MA, Dytfeld D, Grosicki S, Moreau P, Takezako N, Hori M, Leleu X, LeBlanc R, Suzuki K, Raab MS, Richardson PG, Popa McKiver M, Jou YM, Yao D, Das P, San-Miguel J. Elotuzumab Plus Pomalidomide and Dexamethasone for Relapsed/Refractory Multiple Myeloma: Final Overall Survival Analysis From the Randomized Phase II ELOQUENT-3 Trial. J Clin Oncol. 2023 Jan 20;41(3):568-578. doi: 10.1200/JCO.21.02815. Epub 2022 Aug 12. PMID 35960908
- [Derived] Dimopoulos MA, Dytfeld D, Grosicki S, Moreau P, Takezako N, Hori M, Leleu X, LeBlanc R, Suzuki K, Raab MS, Richardson PG, Popa McKiver M, Jou YM, Shelat SG, Robbins M, Rafferty B, San-Miguel J. Elotuzumab plus Pomalidomide and Dexamethasone for Multiple Myeloma. N Engl J Med. 2018 Nov 8;379(19):1811-1822. doi: 10.1056/NEJMoa1805762. PMID 30403938
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 participants were randomized, and 115 participants were treated.
Groups:
- E-Pd Cohort: Elotuzumab + Pomalidomide + Dexamethasone
- Pd Cohort: Pomalidomide + Dexamethasone
Period: Pre-Treatment Period
Arm/Group | E-Pd Cohort | Pd Cohort
Started (Started = Randomized) | 60 | 57
Completed (Completed = Continued into Treatment Period) | 60 | 55
Not Completed | 0 | 2
Not completed — Participant Withdrew Consent | 0 | 2
Period: Treatment Period
Arm/Group | E-Pd Cohort | Pd Cohort
Started | 60 | 55
Completed | 0 | 0
Not Completed | 60 | 55
Not completed — Disease progression | 43 | 38
Not completed — Adverse Event unrelated to study drug | 6 | 9
Not completed — Other reasons | 4 | 2
Not completed — Study drug toxicity | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Maximum Clinical Benefit | 0 | 2
Not completed — Participant request to discontinue | 2 | 0
Not completed — Administrative reasons by sponsor | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Pd Cohort | Pd Cohort | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (9.92) | 65.5 (9.95) | 65.9 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 28 | 22 | 50
    Male | 32 | 35 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 18 | 28
  Unknown or Not Reported | 49 | 39 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    White | 45 | 45 | 90
    Black or African American | 0 | 1 | 1
    Asian | 15 | 9 | 24
    Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of the first documented tumor progression or death due to any cause. Progressive disease response criteria were defined as an increase of 25% from lowest response value in any one or more of the following:
  1. Serum M-component and/or 2. Urine M-component and/or 3. Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels 4. Bone marrow plasma cell percentage; Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia that can be attributed solely to the plasma cell proliferative disorder
Time Frame: From randomization to date of progression or death (up to approximately 21 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | E-Pd Cohort | Pd Cohort
Number analyzed (Participants) | 60 | 57
Months | 10.25 [6.54 to NA] — Upper limit not reached | 4.70 [2.83 to 7.62]
Statistical Analysis 1: Comparison: E-Pd Cohort vs Pd Cohort; Test type: Superiority; p = 0.0043, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.32 to 0.82]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved a best overall response (BOR) of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) using the modified International Myeloma Working Group (IMWG) criteria described as follows, as per investigator's assessment
  * CR: Negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas, and < 5% plasma cells in bone marrow
  * sCR: CR, as defined above, plus the following: Normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  * VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or >= 90% reduction in serum M-protein level plus urine M-protein level < 100 mg per 24 hour
  * PR: >= 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90% or to < 200 mg per 24 hour.
Time Frame: From first dose to disease progression (up to approximately 21 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | E-Pd Cohort | Pd Cohort
Number analyzed (Participants) | 60 | 57
Percent of participants | 58.3 [44.9 to 70.9] | 24.6 [14.1 to 37.8]
Statistical Analysis 1: Comparison: E-Pd Cohort vs Pd Cohort; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.62, 95% CI 2-sided [2.05 to 10.43]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to the date of death from any cause. The survival time for participants who had not died was censored at the last known alive date. OS was censored at the date of randomization for subjects who were randomized but had no follow-up.
Time Frame: From randomization to death (up to approximately 52 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | E-Pd Cohort | Pd Cohort
Number analyzed (Participants) | 60 | 57
Months | 29.80 [22.87 to 45.67] | 17.41 [13.83 to 27.70]
Statistical Analysis 1: Comparison: E-Pd Cohort vs Pd Cohort; Test type: Superiority; p = 0.0217, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.37 to 0.93]

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization to study completion (up to approximately 67 months) SAEs and Other Adverse Events: from first dose to 60 days following last dose (up to approximately 60 months)
Description: All-cause mortality: all randomized participants SAEs and Other Adverse Events: all treated participants
Arm/Group | E-Pd Cohort | Pd Cohort
All-Cause Mortality (participants affected / at risk) | 41/60 | 41/57
Serious Adverse Events (participants affected / at risk) | 42/60 | 33/55
Other Adverse Events (participants affected / at risk) | 56/60 | 49/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-Pd Cohort (N=60) | Pd Cohort (N=55)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 0
Cataract subcapsular (Eye disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Sudden death (General disorders) | 1 | 0
Primary amyloidosis (Immune system disorders) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Pneumococcal sepsis (Infections and infestations) | 2 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pneumonia influenzal (Infections and infestations) | 2 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 3
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 2 | 3
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 7
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-Pd Cohort (N=60) | Pd Cohort (N=55)
Anaemia (Blood and lymphatic system disorders) | 17 | 21
Leukopenia (Blood and lymphatic system disorders) | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 6 | 1
Neutropenia (Blood and lymphatic system disorders) | 16 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 11
Cataract (Eye disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 14 | 6
Diarrhoea (Gastrointestinal disorders) | 15 | 7
Nausea (Gastrointestinal disorders) | 2 | 5
Stomatitis (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 8 | 5
Fatigue (General disorders) | 11 | 8
Oedema peripheral (General disorders) | 11 | 5
Pyrexia (General disorders) | 11 | 12
Bronchitis (Infections and infestations) | 9 | 5
Influenza (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 15 | 9
Oral candidiasis (Infections and infestations) | 1 | 3
Pharyngitis (Infections and infestations) | 5 | 1
Pneumonia (Infections and infestations) | 4 | 3
Respiratory tract infection (Infections and infestations) | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 9
Urinary tract infection (Infections and infestations) | 5 | 3
Blood creatinine increased (Investigations) | 4 | 6
Neutrophil count decreased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 4 | 4
White blood cell count decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 6 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 3
Hypoaesthesia (Nervous system disorders) | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 3
Polyneuropathy (Nervous system disorders) | 4 | 1
Tremor (Nervous system disorders) | 4 | 2
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 6
Hypertension (Vascular disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2015-11-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT02654132/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT02654132/SAP_001.pdf